CLINICAL TRIAL: NCT07217054
Title: Detection of Phosphorylated Alpha-Synuclein in Colonic Tissue Biopsy During Routine Colonoscopy
Brief Title: Colonic Tissue Biopsy Detection of Phosphorylated Alpha-synuclein for Parkinson's Diagnosis or REM Sleep Behavior Disorder
Acronym: Syn-G
Status: Recruiting | Type: Observational
Sponsor: CND Life Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: CND-107
Record Dates: First submitted 2025-10-11; First posted 2025-10-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: PARKINSON DISEASE (Disorder); Parkinson; Parkinson s Disease; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's Disease (PD): Trial participants with Parkinson's disease
- REM Sleep Behavior Disorder (RBD): Trial participants with REM Sleep Behavior Disorder (RBD)

SUMMARY:
The goal of this observational study is to learn whether tissue samples taken from the colon during routine colonoscopy can detect signs of Parkinson's disease or REM Sleep Behavior Disorder (RBD). The main question it aims to answer is:

Can doctors find a protein called alpha-synuclein in colon tissue samples from people with Parkinson's disease and RBD?

Currently, Parkinson's disease is diagnosed by observing symptoms like tremors and movement problems and RBD by loss of muscle atonia during REM sleep, but by then the disease has already progressed significantly. Earlier detection could help doctors start treatment sooner.

DETAILED DESCRIPTION:
What is this study about? This study is testing whether doctors can detect signs of Parkinson's disease or REM Sleep Behavior Disorder (RBD) by taking small tissue samples from the colon during a routine colonoscopy. Researchers want to see if they can find a specific protein called alpha-synuclein that builds up in people with Parkinson's disease or RBD.

Why is this study important? Currently, Parkinson's disease is diagnosed mainly by observing symptoms like tremors and movement problems and RBD is characterized by the loss of muscle atonia during REM sleep. However, by the time these symptoms appear, the disease has already progressed significantly. Finding a way to detect the disease earlier could help doctors start treatment sooner and potentially slow down the disease.

Who can participate?

Adults between 40-99 years old People who have already been diagnosed with Parkinson's disease or REM Sleep Behavior Disorder People who are already scheduled to have a routine colonoscopy for colon cancer screening or other medical reasons What happens during the study?

**During the colonoscopy:**

The colonoscopy procedure remains exactly the same as planned. Doctors will take 4 additional small tissue samples (2 from each side of the colon).

This adds only about 2 minutes to the procedure.

**After the colonoscopy:**

No additional visits are required. The tissue samples will be tested for the alpha-synuclein protein. Participants will not receive individual test results.

What are the risks?

The main risks are the same as any routine colonoscopy, including:

Discomfort during the procedure. Very rare complications like bleeding or bowel perforation. Small risk of infection. Possible breach of medical privacy (researchers take steps to protect this).

What are the benefits?

Participants help advance research that could lead to earlier detection of Parkinson's disease or REM Sleep Behavior Disorder.

This could eventually help future patients get diagnosed and treated sooner. There are no direct medical benefits to participants.

How many people will be in this study? 20 people with Parkinson's disease and 20 people with REM Sleep Behavior Disorder will participate in this study at Digestive Disease Associates (DDA).

How long does participation take?

The colonoscopy procedure (same length as normally planned).

This research is sponsored by CND Life Sciences and conducted at DDA.

ELIGIBILITY:
Inclusion Criteria:

1. Relatively healthy men and women ≥40-99 years of age
2. Patients with a diagnosis of

   1. Clinically confirmed PD or
   2. Clinically confirmed RBD with no diagnosis of PD, DLB or MSA
3. Patients must have agreed to undergo a routine colonoscopy as part of their screening or surveillance for colon cancer or for diagnostic purposes for the exclusion of other GI diseases

Exclusion Criteria:

1. Use of anticoagulants (Plavix or aspirin alone is allowed)
2. Under active treatment for colon cancer; 30-day post anti-cancer treatment allowed
3. Current, ongoing gastrointestinal illness
4. Recent intrabdominal surgery
5. Pregnant or planning to become pregnant before the scheduled colonoscopy
6. Significant cognitive impairment, as determined by study investigators

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with clinically confirmed Parkinson's disease or REM Sleep Behavior Disorder who are undergoing routine colonoscopies for standard medical care. Participants must be able to provide informed consent and understand that participation is voluntary and for research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Detection of phosphorylated alpha-synuclein in colon tissue samples | At time of colonoscopy procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Disease Associates, Branford, Connecticut, United States